CLINICAL TRIAL: NCT05246982
Title: An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) + HLX10 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) + Chemotherapy or HLX07 Monotherapy in Patients With Advanced Metastatic Gastric Cancer
Brief Title: HLX07+HLX10+Chemotherapy or HLX07 Monotherapy in Patients With Advanced Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-GC201
Record Dates: First submitted 2022-02-16; First posted 2022-02-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer (GC) Gastroesophageal Junction Cancer (GEJ)
MeSH Terms: conditions — Stomach Neoplasms | interventions — HLX07

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): HER2 negative and PD-L1 CPS≥5, as first-line therapy
  Interventions: Drug: HLX07+HLX10+oxaliplatin+capecitabine
- Arm B (Experimental): As third-line or above therapy
  Interventions: Drug: HLX07

INTERVENTIONS:
Drug: HLX07+HLX10+oxaliplatin+capecitabine — HLX07 1500mg+HLX10 300mg+oxaliplatin 130mg/m2+capecitabine 1000mg/m2 q3w
  Arms: Arm A
Drug: HLX07 — HLX07 1500mg q3w
  Arms: Arm B

SUMMARY:
This study is conducted in patients with advanced metastatic gastric cancer including gastroesophageal junction cancer. This study includes two arms: A and B. Arm A (patients with HER2 negative and PD-L1 CPS≥5 ) will receive HLX07 combination therapy with HLX10 and chemotherapy (oxaliplatin+capecitabine) as first-line treatment. Arm B will receive HLX07 monotherapy as third-line or above treatment. All of eligible patients will receive study drug treatment until loss of clinical benefit, unacceptable toxicity, death, withdrawal of informed consent (whichever occurs first, HLX10 treatment up to 2 years).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF); be willing to follow and be able to complete all study procedures;
2. Age ≥ 18 years and ≤ 75 years when ICF is signed;
3. Unresectable locally advanced, or metastatic gastric cancer including gastroesophageal junction cancer, and histopathologically confirmed diagnosis of adenocarcinoma;
4. Arm A: never received systemic anti-tumor drug therapy before, with HER2 negative and PD-L1 CPS≥5; Arm B: failed to prior systemic anti-tumor therapy (at least 2 lines);
5. Measurable lesion according to RECIST v1.1 by IRRC;
6. ECOG score 0-1;
7. Expected survival 12 weeks.

Exclusion Criteria:

1. Has other active malignancies within 5 years before the first administration of the study drug;
2. Plan to or have previously received organ or bone marrow transplantation;
3. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
4. Arm A: previously received antibody drugs against immune checkpoints (such as PD-1, PD-L1, CTLA4, etc.) and / or antibody drugs against EGFR; Arm B: previously received antibody drug treatment against EGFR;
5. Have received any research drugs within 14 days before the first use of the study drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 2 years
  Objective response rate by IRRC assessment per RECIST 1.1
PFS | From the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier), assessed up to 2 years
  Progression-free survival by IRRC assessment per RECIST 1.1

SECONDARY OUTCOMES:
OS | From the date of first dose unitl the date of death from any cause，assessed up to 2 years
  Overall survival
ORR | Up to 2 years
  Objective response rate by INV assessment per RECIST 1.1
PFS | From the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier), assessed up to 2 years
  Objective response rate by INV assessment per RECIST 1.1
DOR | From the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response by IRRC/INV assessment per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Gansu Wuwei Tumor Hospital, Wuwei, Gansu
  - Fudan University shanghai cancer center, Shanghai